CLINICAL TRIAL: NCT00889720
Title: A Multicenter, Open Label Study To Investigate The Feasibility And Efficacy Of A Smoking Cessation Program With Varenicline In Patients Undergoing Elective Surgery
Brief Title: A Pilot Study Of Smoking Cessation Treatment Including Varenicline In Patients Scheduled For Planned Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A3051113
Record Dates: First submitted 2009-04-28; First posted 2009-04-29 (Estimated); Results first posted 2011-08-25 (Estimated); Last update posted 2011-10-17 (Estimated); Status verified 2011-07

CONDITIONS: Smoking Cessation
Keywords: smoking cessation; varenicline; elective surgery; wound infections; post-operative complications
MeSH Terms: conditions — Smoking Cessation; Wound Infection | interventions — Varenicline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Smoking cessation tratment including varenicline (Other)
  Interventions: Drug: Varenicline

INTERVENTIONS:
Drug: Varenicline — Varenicline film coated tablets - escalating dose with maximum dose of 1mg bd
  Other Names: Champix

SUMMARY:
It is possible to offer smoking cessation treatment including varenicline to patients scheduled for elective surgery. This study will evaluate whether or not this will enable some patients to quit smoking for up to 4 weeks prior to surgery and in turn, whether this may lead to reductions in post-operative complication such as wound infections.

DETAILED DESCRIPTION:
Recruitment to this study was terminated (on February 23, 2010) earlier than originally planned because recruitment was much slower than expected and therefore the study has already achieved its main objective of assessing the feasibility of conducting a larger study of similar design to investigate the efficacy of smoking cessation therapy in a pre-surgical setting. The decision to end recruitment to the trial was not based on any safety concerns.

ELIGIBILITY:
Inclusion Criteria:

* Smokers motivated to stop smoking scheduled for elective surgery

Exclusion Criteria:

* Current or recent depression
* Current or recent suicidal ideation
* Uncontrolled or unstable clinically significant medical condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-11; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- Pfizer Investigational Site, Paris, France
- Pfizer Investigational Site, Pisa, Italy

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3051113&StudyName=A%20Pilot%20Study%20Of%20Smoking%20Cessation%20Treatment%20Including%20Varenicline%20In%20Patients%20Scheduled%20For%20Planned%20Surgery

RESULTS

PARTICIPANT FLOW:
Groups:
- Varenicline: Week 1: Day 1 through Day 3: varenicline 0.5 mg once a day, Day 4 through Day 7: varenicline 0.5 mg twice daily (BID); Week 2 through Week 12: varenicline 1 mg BID with option to reduce to 0.5 mg BID depending on toleration.
Period: Overall Study
Arm/Group | Varenicline
Started | 16
Surgical Population | 12
Completed | 8
Not Completed | 8
Not completed — Withdrawal by Subject | 4
Not completed — Other | 4

BASELINE CHARACTERISTICS:
Arm/Group | Varenicline
Number analyzed (Participants) | 16
Age, Customized [Number; unit: Participants]
  Between 18 and 44 years | 6
  Between 45 and 64 years | 7
  >= 65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 9

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Fully Compliant Participants
Description: Compliance defined as completed 12 weeks of varenicline therapy, underwent surgery 8 weeks +-10 days after start of varenicline treatment, and had evaluations of wound infection 1 to 3 days and 6 to 10 days after surgery.
Time Frame: Baseline through Week 12
Population: Surgical Population: subset of Full Analysis Set; includes all participants who took at least 1 dose (including partial doses) of study medication and received their planned surgery within the study period. N = participants in surgical population.
Measure: Number; unit: percentage of participants
Arm/Group | Varenicline
Number analyzed (Participants) | 12
percentage of participants | 0

2. Primary Outcome: Number of Participants With Surgical Site Infection Post-surgery Days 1 to 3: Center for Disease Control (CDC) Definition
Description: Surgical site infections (SSIs) assessed by 1992 CDC definition; divided into incisional and organ/space SSIs. Incisional space SSIs further classified as involving only skin and subcutaneous tissue (superficial incisional) or involving deep soft tissues (fascial and muscle layers) of the incision (deep incisional ). Organ/space SSIs involve any part of the anatomy (organs or spaces) other than incision opened or manipulated during operative procedure. None = did not have a surgical site infection. Category 0 = no surgical wound complications. Not done = not assessed.
Time Frame: Post-surgery Days 1-3
Population: Surgical Population; N= number of participants with a Day 1-3 post-surgery visit.
Measure: Number; unit: participants
Arm/Group | Varenicline
Number analyzed (Participants) | 12
participants
  Category 0: no surgical wound complications | 11
  Not done | 1

3. Primary Outcome: Number of Participants With Surgical Site Infection Post-surgery Days 6 to 10: Center for Disease Control (CDC) Definition
Description: as for outcome 2
Time Frame: Post-surgery Days 6-10
Population: Surgical Population; N= number of participants with a Day 6-10 post-surgery visit.
Measure: Number; unit: participants
Arm/Group | Varenicline
Number analyzed (Participants) | 12
participants
  Category 0: no surgical wound complications | 11
  Not Done | 1

4. Primary Outcome: Number of Participants With Surgical Site Infection at Week 12: Center for Disease Control (CDC) Definition
Description: as for outcome 2
Time Frame: Week 12
Population: Surgical Population; N= number of participants with a Week 12 visit.
Measure: Number; unit: participants
Arm/Group | Varenicline
Number analyzed (Participants) | 11
participants
  Category 0: no surgical wound complications | 9
  Not done | 2

5. Primary Outcome: Number of Participants With Surgical Site Infection at Week 26: Center for Disease Control (CDC) Definition
Description: as for outcome 2
Time Frame: Week 26
Population: Surgical Population; N= number of participants with a Week 26 visit.
Measure: Number; unit: participants
Arm/Group | Varenicline
Number analyzed (Participants) | 9
participants
  Category 0: no surgical wound complications | 9
  Not done | 0

6. Primary Outcome: Number of Participants With Surgical Site Infections With Microbiological Confirmation of Bacterial Infection
Description: Microbiological confirmation defined as organisms isolated from an aseptically obtained culture of fluid or tissues from the superficial incision.
Time Frame: Post-surgery Days 1-3, Post-surgery Days 6-10, Week 12, Week 26
Population: Surgical Population; Due to satisfactory wound healing in all subjects, microbiological assessment was not necessary and no swabs were taken.
Measure: Number; unit: participants
Arm/Group | Varenicline
Number analyzed (Participants) | 0

7. Primary Outcome: Number of Participants With Grade of Wound Healing and Severity of Surgical Site Infections Post-surgery Days 1 to 3: Southampton Wound Assessment Scale
Description: Grade 0 = normal healing (NH); Grade I = NH with (w) mild bruising (br) or haematoma (a: some br, b: considerable br, c: mild erythema); Grade II= erythema plus other signs of inflammation (a: at 1 point, b: around sutures, c: along wnd, d: around wnd); Grade III= clear or haemoserous discharge (a: at 1 point only ≤ 2 cm, b: along wnd > 2 cm, c: large volume, D: prolonged > 3 days); Grade IV= pus (a: at 1 point only ≤ 2 cm, b: along wnd > 2 cm; Grade V=deep or severe wnd infection (w or without tissue breakdown; haematoma requiring aspiration). Not done = not assessed.
Time Frame: Post-surgery Days 1-3
Population: Surgical Population; N= number of participants with a Day 1-3 post-surgery visit.
Measure: Number; unit: participants
Arm/Group | Varenicline
Number analyzed (Participants) | 12
participants
  Grade 0 | 10
  Grade Ia | 1
  Not done | 1

8. Primary Outcome: Number of Participants With Grade of Wound Healing and Severity of Surgical Site Infections Post-surgery Days 6 to 10: Southampton Wound Assessment Scale
Description: as for outcome 7
Time Frame: Post-surgery Days 6-10
Population: Surgical Population; N= number of participants with a Day 6-10 post-surgery visit.
Measure: Number; unit: participants
Arm/Group | Varenicline
Number analyzed (Participants) | 12
participants
  Grade 0 | 8
  Grade Ia | 1
  Grade IIa | 1
  Grade IIb | 1
  Not done | 1

9. Primary Outcome: Number of Participants With Grade of Wound Healing and Severity of Surgical Site Infections at Week 12: Southampton Wound Assessment Scale
Description: as for outcome 7
Time Frame: Week 12
Population: Surgical Population; N= number of participants with a Week 12 visit.
Measure: Number; unit: participants
Arm/Group | Varenicline
Number analyzed (Participants) | 11
participants
  Grade 0 | 8
  Grade Ia | 1
  Not done | 2

10. Primary Outcome: Number of Participants With Grade of Wound Healing and Severity of Surgical Site Infections at Week 26: Southampton Wound Assessment Scale
Description: as for outcome 7
Time Frame: Week 26
Population: Surgical Population; N= number of participants with a Week 26 visit.
Measure: Number; unit: participants
Arm/Group | Varenicline
Number analyzed (Participants) | 9
participants
  Grade 0 | 8
  Not done | 1

11. Primary Outcome: Wound Healing Grade by ASEPSIS Criteria: Post-surgery Days 1 to 3
Description: Wound grading scale of wound characteristics assessed by portion of wound infected and point scale for daily wound inspection. Infections categorized by ASEPSIS score as satisfactory healing (0-10), disturbance of healing (11-20), minor wound infection (21-30), moderate wound infection (31-40), and severe wound infection (>40). Surgical site complication defined as total score >10; wound infection defined as total score >20. Not done = not assessed.
Time Frame: Post-surgery Days 1-3
Population: Surgical Population; N= number of participants who had ASEPSIS wound grading during the study and had a Day 1-3 post-surgery visit.
Measure: Number; unit: participants
Arm/Group | Varenicline
Number analyzed (Participants) | 8
participants
  Satisfactory healing | 7
  Not done | 1

12. Primary Outcome: Wound Healing Grade by ASEPSIS Criteria: Post-surgery Days 6 to 10
Description: as for outcome 11
Time Frame: Post-surgery Days 6-10
Population: Surgical Population; N= number of participants who had ASEPSIS wound grading during the study and had a Day 6-10 post-surgery visit.
Measure: Number; unit: participants
Arm/Group | Varenicline
Number analyzed (Participants) | 8
participants
  Satisfactory healing | 7
  Not done | 1

13. Primary Outcome: Wound Healing Grade by ASEPSIS Criteria at Week 12
Description: as for outcome 11
Time Frame: Week 12
Population: Surgical Population; N = number of participants who had ASEPSIS wound grading during the study and had a Week 12 visit.
Measure: Number; unit: participants
Arm/Group | Varenicline
Number analyzed (Participants) | 7
participants
  Satisfactory healing | 6
  Not done | 1

14. Primary Outcome: Wound Healing Grade by ASEPSIS Criteria at Week 26
Description: as for outcome 11
Time Frame: Week 26
Population: Surgical Population; N = number of participants who had ASEPSIS wound grading during the study and had a Week 24 visit.
Measure: Number; unit: participants
Arm/Group | Varenicline
Number analyzed (Participants) | 6
participants
  Satisfactory healing | 6
  Not done | 0

15. Primary Outcome: Number of Participants With 7 Day Point Prevalence (PP) for Smoking Abstinence Prior to Hospital Admission.
Description: Responder defined as participant who answered "No" to question on Nicotine Use Inventory (NUI), "Has the subject smoked any cigarettes or cigarillos or used any other nicotine containing products in the last 7 days?" Additionally, responder status confirmed by measurement of end-expiratory exhaled carbon monoxide concentration <10 parts per million (ppm).
Time Frame: 7 days prior to hospital admission to day of hospital admission (after Week 8 of treatment)
Population: Surgical population: N = participants who took at least 1 dose of study medication and received planned surgery.
Measure: Number; unit: participants
Arm/Group | Varenicline
Number analyzed (Participants) | 12
participants | 9

16. Secondary Outcome: Number of Participants by Severity of Post-operative Complications: Dindo, Demartines and Clavien Classification System
Description: Grade 0: no post-operative (post-op) complications (comp), Grade 1: any deviation from normal post-op course without need for pharmacological treatment (PT) other than allowed interventions (INT), or surgical, endoscopic or radiological INT; Grade II: required PT with drugs other than those allowed for grade I comp; Grade III required surgical, endoscopic or radiological INT, IIIa: not under general anaesthesia (GA), IIIb: under GA; Grade IV: life-threatening comp requiring IC/ICU management, IVa: single organ dysfunction (DSF), IVb: multiorgan DSF; Grade V: death. Not done = not assessed.
Time Frame: Baseline through Week 26
Population: Surgical Population; N = participants who took at least 1 dose of study medication and received planned surgery. Results provided for participants who had a study visit at timepoint. For participants with more than 1 incidence of surgical complication recorded, the most severe incidence was used for analysis. Abbreviations: PS=post-surgery.
Measure: Number; unit: participants
Arm/Group | Varenicline
Number analyzed (Participants) | 12
participants
  1-3 days PS: No post-operative complications | 10
  1-3 days PS: Grade II | 1
  1-3 days PS: Not done | 1
  6-10 days PS: No post-operative complications | 7
  6-10 days PS: Grade I | 3
  6-10 days PS: Grade II | 1
  6-10 days PS: Not done | 1
  Week 12: No post-operative complications | 7
  Week 12: Grade II | 1
  Week 12: Grade IIIb | 1
  Week 12: Not done | 2
  Week 26: No post-operative complications | 8
  Week 26: Grade IIIb | 1

17. Secondary Outcome: Percentage of Participants Who Succeed in Reducing Their Cigarette Consumption by at Least 50% in 7 Days Preceding Hospital Admission Compared With Baseline.
Time Frame: Baseline, Week 8
Population: Surgical population. Not analyzed due the limited number of participants recruited.
Measure: Number; unit: percentage of participants
Arm/Group | Varenicline
Number analyzed (Participants) | 0

18. Secondary Outcome: Number of Participants With 7-day Point Prevalence (PP) for Abstinence From Cigarette Smoking and Other Nicotine Use at the End of Treatment (Week 12)
Description: as for outcome 15
Time Frame: Week 12
Population: Surgical population: N = number of participants who had a Week 12 visit.
Measure: Number; unit: participants
Arm/Group | Varenicline
Number analyzed (Participants) | 11
participants | 9

19. Secondary Outcome: Number of Participants With 7 Day Point Prevalence (PP) for Abstinence in the Week Preceding Week 26
Description: as for outcome 15
Time Frame: Week 26
Population: Surgical population: N = number of participants who had a Week 26 visit.
Measure: Number; unit: participants
Arm/Group | Varenicline
Number analyzed (Participants) | 9
participants | 7

20. Secondary Outcome: Percentage of Participants Who Reduced Their Cigarette Consumption by at Least 50% in the 7 Days Preceding Weeks 12 and 26 Compared With Baseline.
Time Frame: Baseline, Week 12, Week 26
Population: Surgical population: Not analyzed due the limited number of participants recruited.
Measure: Number; unit: percentage of participants
Arm/Group | Varenicline
Number analyzed (Participants) | 0

21. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events by Type, Severity, Seriousness, and Relatedness to Varenicline
Description: Treatment-emergent AE (TEAE): any untoward medical occurrence that occurred or worsened after beginning study treatment without regard to causal relationship. Treatment-related TEAE: investigator assessment of reasonable possibility that treatment caused or contributed to AE. Severe TEAE: interfered significantly with usual function. SAE: AE resulting in death, initial or prolonged inpatient hospitalization, a life-threatening experience (immediate risk of death), persistent or significant disability/incapacity, congenital anomaly, or deemed significant for any other reason.
Time Frame: Baseline through Week 26 (within 30 days of last dose)
Population: Safety analysis set: participants who took at least 1 dose (including partial doses) of study medication. N = number of treated subjects. Includes data up to 30 days after last dose of study drug.
Measure: Number; unit: participants
Arm/Group | Varenicline
Number analyzed (Participants) | 16
participants
  TEAE: all causalities | 9
  TEAE: treatment-related | 8
  Severe TEAE: all causalities | 3
  Severe TEAE: treatment-related | 1
  SAE: all causalities | 1
  SAE: treatment-related | 0

22. Secondary Outcome: Number of Treatment Emergent Adverse Events by Severity
Description: Mild: did not interfere with usual function; Moderate: interfered to some extent with usual function; Severe: interfered significantly with usual function. If the same participant in a given treatment had more than one occurrence in the same preferred term event category, only the most severe occurrence was taken. Missing baseline severities were imputed as mild.
Time Frame: Baseline through Week 26 (within 30 days of last dose)
Population: Safety analysis set. N = number of treated subjects. Includes data up to 30 days after last dose of study drug.
Measure: Number; unit: events
Arm/Group | Varenicline
Number analyzed (Participants) | 16
events
  Mild | 13
  Moderate | 11
  Severe | 4

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Varenicline
Serious Adverse Events (participants affected / at risk) | 1/16
Other Adverse Events (participants affected / at risk) | 9/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Varenicline (N=16)
Intestinal obstruction (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Varenicline (N=16)
Tachycardia (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 2
Asthenia (General disorders) | 1
Feeling abnormal (General disorders) | 1
Gastroenteritis (Infections and infestations) | 1
Viral rhinitis (Infections and infestations) | 1
Incision site pain (Injury, poisoning and procedural complications) | 1
Transaminases increased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Abnormal dreams (Psychiatric disorders) | 1
Decreased interest (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 3
Libido decreased (Psychiatric disorders) | 1
Mental disorder (Psychiatric disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension (Vascular disorders) | 1
Lymphoedema (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
This study was terminated after 16 of 100 planned subjects were enrolled due to slow recruitment and non-compliance with the protocol; only selected efficacy listings of the surgical population and key safety data were reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.